CLINICAL TRIAL: NCT06899243
Title: The Effect of CL22205 on Bone Mineral Density and Menopausal Symptoms in Women: A Randomized, Double-blind, Placebo Controlled Clinical Trial
Brief Title: Efficacy of CL22205 on Bone Mineral Density and Menopausal Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eetho Brands, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EB/MS/CL22205/24
Record Dates: First submitted 2025-03-01; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Menopausal Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL22205 (Experimental): 200 mg, One capsule a day after breakfast for 360 days
  Interventions: Dietary Supplement: CL22205
- Placebo (Other): One capsule a day after breakfast for 360 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CL22205 — 200 mg, Route : Oral, One capsule a day after breakfast for 360 days
  Arms: CL22205
Other: Placebo — Route : Oral, One capsule a day after breakfast for 360 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of CL22205 on bone mineral density and menopausal symptoms in women.

DETAILED DESCRIPTION:
A total of 80 healthy female subjects aged between 55 and 65 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either CL22205 - 200 mg or placebo arms at 1:1 ratio. The subjects will be instructed to take one capsule a day after breakfast for 360 days. Apart from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition's safety and tolerability. The safety assessment of the CL22205 will also include routine laboratory investigations on blood, urine and clinical chemistry at screening and the final visit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females aged between 55 and 65 years with a Body mass index (BMI) of approximately 24 and 29 kg/m2.
* Women with menopausal symptoms (modified Kupperman index scores 15-29), absence of menstrual cycle for past 12-months; follicle-stimulating hormone (FSH) > 30 mIU/mL; estradiol < 30 pg/mL.
* Subjects who are under standard supplementation of Vitamin D3 (cholecalciferol) and calcium carbonate.
* Subjects with osteopenia (T score of spine between -1 and -2.5 in DEXA).
* Must also be experiencing at least two symptoms of menopause, such as sleep disturbances, mood changes, fatigue and lack of energy, changes in sexual function, urinary changes, weight gain, or vaginal changes.
* Subject understands the study procedures and provides signed informed consent to participate in the study.
* Normal vital signs, including electrocardiogram (ECG) and laboratory evaluations (including clinical biochemistry, haematology, lipid profile, thyroid profile and complete urinalysis) within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.

Exclusion Criteria:

* Consumption of functional food or supplement that modifies body composition, during or 6 months prior to the study.
* History of cerebrovascular disease, thrombo-embolic disorders, heart attack, or angina at any time or thrombophlebitis within the last 5 years.
* Subjects on anti-coagulant or anti-platelet drugs on a daily basis for any conditions.
* Presence of chronic diseases that prevent the performance of a physical exercise program (disabling arthropathies, moderate / severe chronic lung disease, arrhythmias, etc.).
* High alcohol intake (>2 standard drinks per day), or recreational drugs (such as cocaine, methamphetamine, marijuana, etc.) or psychiatric drug users.
* Smokers or tobacco users.
* Inability to understand informed consent.
* Serious or terminal illnesses.
* Fasting blood glucose level >125 mg/dl.
* Subjects with a high blood pressure at screening (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg).
* Subjects who had any hormonal therapy, metformin or any other herbal products in the past 3 months.
* Hypothyroidism, hyperthyroidism, hyperprolactinemia, Cushing's syndrome and congenital adrenal hyperplasia, following a special diet for the past 3 months.
* Taking drugs affecting insulin sensitivity or lipid and hormonal profiles, including glucocorticoids, ovulation-stimulating drugs, anti-obesity, anti-diabetes, anti-hypertensive, anti-estrogenic, anti-androgenic during the last 3 months (except the usual drugs of the subjects).
* Active gall bladder disease, gynaecological (including hysterectomy) or breast surgery in the last 6 months.
* Subjects who are being treated for liver cancer or cirrhosis, chronic renal failure, congestive heart failure.
* Subjects with a systemic disease including tuberculosis, leucosis, collagenosis, multiple sclerosis or other autoimmune diseases.
* History of breast, endometrial, other gynaecological cancer at any time or other cancer within the last 5 years.
* History of hypersensitivity reactions attributed to investigational product (IP) or its components or related products.
* History of positive hepatitis screening including Hepatitis B surface antigen or Hepatitis C virus (HCV) antibodies or subjects with human immunodeficiency virus (HIV) and /or syphilis.
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
* Participated in a clinical study with an investigational drug or biologic within the last 30 days.
* Any condition that in opinion of the investigator, does not justify the subjects' participation in the study.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy females with Menopausal symptoms
Enrollment: 80 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in : Bone Mineral density (BMD) (g/cm2) of Lumbar spine (L1-L4) | Screening/Baseline, Days 180 & 360
  A low-dose X-ray is used to assess the bone mineral content (density) in specific areas, such as the lumbar spine at L1-L4 region. The results are typically expressed in terms of the T-score. If T scores ≥-1 signifies healthy bone, a range from -1 to -2.5 indicates osteopenia and a score of ≤-2.5 indicates osteoporosis.

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in : Lean body mass through DEXA | Screening/Baseline, Days 180 & 360
  Dual-energy X-ray absorptiometry (DEXA) uses two X-ray beams with different energies to measure lean body mass in Kilograms. Higher ranges reflect a greater proportion of lean tissue.
Change from baseline to the end of the study period in : Scores of modified Kupperman index (mKI) | Screening, Baseline/Day 1, Days 90,180 & 360
  The modified Kupperman Index (mKI) is a tool used to assess the severity of menopausal symptoms. The total score ranges from 0 to 63, calculated as the sum of all items by the weighting factor. Scores ranging from 0-6, 7-15, 16-30, and >30 were used to rate the degree of severity as none, mild, moderate, and severe, respectively.
Change from baseline to the end of the study period in: Hand grip-strength | Baseline/Day 1, Days 90,180 & 360
  Grip strength was a measure of muscular strength (in kgs) or the maximum force/tension generated by one's forearm muscles. The Hand grip strength was measured using digital hand dynamometer.
Change from baseline to the end of the study period in: Chalder Fatigue Scale (CFS) | Baseline/Day 1, Days 90,180 & 360
  The Fatigue Scale, sometimes referred to as the Chalder Fatigue Scale, is a self-administered questionnaire for measuring the extent and severity of fatigue within both clinical and non-clinical, epidemiological populations. Items are rated on a 4-point Likert scale (0, 1, 2, 3), with higher scores indicating greater fatigue. The respondent's global score can range from 0 to 33.
Change from baseline to the end of the study period in: Profile of Mood States (POMS-SF) | Baseline/Day 1, Days 90,180 & 360
  POMS-SF is a commonly used tool for examining people's emotional states. The total score ranges from 0 to 100. A Total Mood Disturbance (TMD)is calculated by subtracting the vigour score from the total sum of the raw scores for tension, depression, anger, fatigue, and confusion. The lower scores indicative of people with more stable mood profiles.
Change from baseline to the end of the study period in: Female Sexual Function Index (FSFI) | Baseline/Day 1, Days 90,180 & 360
  The FSFI was developed as a brief, easy-to-administer, self-report tool for assessing key dimensions or domains of sexual function and quality of life in various populations of women. Female Sexual Function Index (FSFI), a widely used tool with six domains (Arousal, Desire, Orgasm, Lubrication, Satisfaction, and Pain). The total FSFI score ranges from minimum score of 2 and maximum score of 36. Greater Scores indicates better sexual function.
Change from baseline to the end of the study period in: Pittsburgh Sleep Quality Index (PSQI) | Baseline/Day 1, Days 90,180 & 360
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, global PSQI score range of 0-21, with higher scores indicating more acute sleep disturbances.
Change from baseline to the end of the study period in : Menopause Symptoms' Severity Inventory (MSSI-38) | Baseline/Day 1, Days 90,180 & 360
  The Menopause Symptoms' Severity Inventory (MSSI-38) is a comprehensive tool used to assess menopausal symptoms in terms of both frequency and intensity. MSSI-38 is scored using a five-point Likert scale. The total score ranges from 0 to 152. As the score increases, severity and intensity of menopausal symptoms increases.
Change from baseline to the end of the study period in : Mini Cog Questionnaire (Cognitive function) | Baseline/Day 1, Days 90,180 & 360
  The Mini-Cog was one such neuropsychological test that has been effective in detecting patients with dementia. It consists of a three-item recall test and a clock drawing test (CDT). For the three-recall score, ranges from 0-3, and in CDT, subjects were asked to spontaneously draw a circular clock displaying a particular time (11:10). 2 points for a normal clock or 0 (zero) points for an abnormal clock drawing (Lowest possible Score: 0 and the highest possible score: 5). The 3-item recall and clock drawing scores were added together to get the final score. Scores ranges from 0-5, with an increase in score reflect an improvement in cognitive function.
Change from baseline to the end of the study period in : Subject's self-assessment of skin Questionnaire | Baseline/Day 1, Days 90,180 & 360
  As the perception of the skin radiance is subjective, a self-assessment has been performed through a questionnaire. The scores range from 0 to 10, with higher scores indicating better skin quality in terms of complexion, smoothness, texture, elasticity, and hydration.
Change from baseline to the end of the study period in : Scores of subjective self-assessment on hair quality | Baseline/Day 1, Days 90,180 & 360
  This is a subjective measurement of hair quality by considering the hair fall rate. The Highest Possible Score is 5.
Change from baseline to the end of the study period in : Nail quality related questionnaire (NailQoL) | Baseline/Day 1, Days 90,180 & 360
  The Nail Quality of Life (NailQOL) is a measure or assessment used to evaluate how nail condition (such as nail diseases or abnormalities) impacts an individual overall quality of life. NailQOL of 15 questions will be administered and each question will be scored on a 0-100 scale, where 0 = never; 25 = rarely; 50 = sometimes; 75 = often; 100 = all the time. The average total score ranges between 0 and 100. An increase in Nail QoL scores indicates worsening quality of life.
Change from baseline to the end of the study period in : Gastrointestinal symptoms questionnaire (GIS) | Baseline/Day 1, Days 90,180 & 360
  GIS questionnaire includes questions about the severity of GI symptoms (Abdominal pain, Epigastric pain, general intestinal symptoms, dysphagia, and stools). The total highest possible Score is 30 and the total lowest possible score is 0.
Change from baseline to the end of the study period in : Perceived Stress Scale (PSS-10) | Baseline/Day 1, Days 90,180 & 360
  The perceived stress scale (PSS) is the most widely used psychological questionnaire containing ten questions for measuring the perception of stress. The total highest possible Score is 30 and the total lowest possible score is 0.
Change from baseline to the end of the study period in : Visual assessment of skin wrinkles | Baseline/Day 1, Days 90,180 & 360
  Visual assessment of skin wrinkles used to evaluate the appearance of skin aging and to determine the severity of wrinkles. This kind of assessment is typically done by a healthcare professional or dermatologist and involves examining the skin surface to identify and score wrinkles. Grade ranging from 0 to 9 where 0 represents no wrinkles and 9 represents deep wrinkles.
Change from baseline to the end of the study period in : Core Lower Urinary Tract Symptom score (CLSS) | Baseline/Day 1, Days 90,180 & 360
  The core lower urinary tract symptom score (CLSS) questionnaire addresses 10 important lower urinary tract symptoms, which are reported as the most influential symptoms that have a negative impact on the QoL of symptomatic men and women. The total score ranges between 0 and 30. Higher scores reflect greater symptom severity.
Change from baseline to the end of the study period in: Vaginal pH | Baseline/Day 1, Days 90,180 & 360
  The vaginal pH was assessed by using a pH test strip.
Change from baseline to the end of the study period in : Skin hydration using moisture meter | Baseline/Day 1, Days 90,180 & 360
  Skin hydration means the moisture content present on the surface of the skin. This will be done by using a moisture meter.
Change from baseline to the end of the study period in : Bone specific serum ALP | Baseline/Day 1 & Day 360
  Bone-specific ALP, produced by osteoblasts, is an enzyme vital for bone mineralization. It's a marker for bone formation and turnover, with elevated levels indicating increased bone formation (e.g., Paget's disease) and decreased levels indicating reduced bone formation (e.g., osteoporosis).
Change from baseline to the end of the study period in : Serum Osteoprotegerin | Baseline/Day 1 & Day 360
  Osteoprotegerin (OPG), produced by osteoblasts, is a key regulator of bone resorption. It inhibits osteoclast differentiation and activity, thereby influencing bone density. OPG also plays a role in vascular calcification and cardiovascular disease. As a marker of bone turnover, elevated OPG levels are associated with increased bone density (e.g., osteopetrosis, Paget's disease), while decreased levels correlate with reduced bone density, osteoporosis, and increased fracture risk.
Change from baseline to the end of the study period in : Serum Osteocalcin | Baseline/Day 1 & Day 360
  Osteocalcin, a protein hormone secreted by osteoblasts, is fundamental to bone mineralization and calcium homeostasis. It promotes calcium deposition, modulates bone resorption, and participates in glucose metabolism and fat mass regulation. As a biomarker of bone formation, elevated osteocalcin levels indicate increased bone turnover (e.g., osteoporosis, Paget's disease), while decreased levels suggest reduced bone formation (e.g., osteomalacia, rickets).
Change from baseline to the end of the study period in: Serum cortisol | Baseline/Day 1 & Day 360
  Cortisol, a steroid hormone synthesized by the adrenal glands, is essential for the body's stress response, glucose regulation, and macronutrient metabolism. Maintaining appropriate cortisol levels is critical for women's overall health.
Change from baseline to the end of the study period in: Vaginal dryness | Baseline/Day 1, Days 90,180 & 360
  The vaginal dryness intensity was assessed with an analog visual scale (length 10 cm), considering 10 as the maximum vaginal dryness and 0 as symptom absence.

OTHER OUTCOMES:
Telephonic evaluation: Modified Kupperman index (mKI) | Monthly (Every month between evaluation days)
  The modified Kupperman Index is a tool used to assess the severity of menopausal symptoms. The total score ranges from 0 to 63, with scores of 0-6, 7-15, 16-30, and over 30 used to classify the severity as none, mild, moderate, and severe, respectively.
Telephonic evaluation: Chalder Fatigue Scale (CFS) | Monthly (Every month between evaluation days)
  Chalder Fatigue Scale is used to measuring the extent and severity of fatigue. Items are rated on a 4-point Likert scale (0, 1, 2, 3), with higher scores indicating greater fatigue. The respondent's global score can range from 0 to 33.
Telephonic evaluation: Female Sexual Function Index (FSFI) | Monthly (Every month between evaluation days)
  The Female Sexual Function Index was developed for assessing key dimensions or domains of sexual function and quality of life in women. The total FSFI score ranges from 2 to 36. Greater Scores indicates better sexual function.
Telephonic evaluation: Pittsburgh Sleep Quality Index (PSQI) | Monthly (Every month between evaluation days)
  The Pittsburgh Sleep Quality Index is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Global PSQI score range of 0-21, with higher scores indicating more acute sleep disturbances.
Telephonic evaluation: Profile of Mood States (POMS-SF) | Monthly (Every month between evaluation days)
  Profile of Mood States is a commonly used tool for examining people's emotional states. The total score ranges from 0 to 100. The lower scores are indicative of people with more stable mood profiles.
Telephonic evaluation: Menopause Symptoms' Severity Inventory (MSSI-38): | Monthly (Every month between evaluation days)
  The Menopause Symptoms' Severity Inventory is a comprehensive tool used to assess menopausal symptoms in terms of both frequency and intensity. The total score ranges from 0 to 152. As the score increases, severity and intensity of menopausal symptoms increases.
Telephonic evaluation: Subject's self-assessment of skin questionnaire | Monthly (Every month between evaluation days)
  As the perception of the skin radiance is subjective, a self-assessment has been performed through a questionnaire. The score ranges from 0to 10, with higher scores indicating better skin quality in terms of complexion, smoothness, texture, elasticity, and hydration.
Telephonic evaluation: Scores of subjective self-assessments on hair quality | Monthly (Every month between evaluation days)
  This is a subjective measurement of hair quality by considering the hair fall rate. The Highest Possible Score is 5.
Telephonic evaluation: Nail quality related questionnaire (NailQoL) | Monthly (Every month between evaluation days)
  The Nail Quality of Life is a measure or assessment used to evaluate how nail condition (such as nail diseases or abnormalities) impacts an individual overall quality of life. Na of 15 questions will be administered, and each question will be scored on a 0-100 scale, where 0 = never; 25 = rarely; 50 = sometimes; 75 = often; 100 = all the time. The average total score ranges between 0 and 100. An increase in Nail QoL scores indicates worsening quality of life.
Telephonic evaluation: Core Lower Urinary Tract Symptom score (CLSS) | Monthly (Every month between evaluation days)
  The core lower urinary tract symptom score questionnaire addresses 10 important lower urinary tract symptoms. The total score ranges between 0 and 30. Higher scores reflect greater symptom severity.
Telephonic evaluation: Perceived Stress Scale (PSS-10) | Monthly (Every month between evaluation days)
  The perceived stress scale is the most widely used psychological questionnaire containing ten questions for measuring the perception of stress. The total highest possible score is 30 and the total lowest possible score is 0.
Telephonic evaluation: Gastrointestinal symptoms questionnaire (GIS) | Monthly (Every month between evaluation days)
  Gastrointestinal symptoms questionnaire includes questions about the severity of GI symptoms (Abdominal pain, Epigastric pain, general intestinal symptoms, dysphagia, and stools). The total highest possible Score is 30 and the total lowest possible score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Arti Dibya, MBBS, MS DGO, Principal Investigator — Vastalya Hospital and multispecialty Centre

IPD SHARING:
Plan to Share IPD: No